CLINICAL TRIAL: NCT00555022
Title: A Randomized Double-blind, Placebo-controlled, Crossover, Dose Escalation Study to Examine the Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of Single Inhaled Doses of GSK1160724 and Tiotropium Bromide
Brief Title: Effect of GSK1160724 In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: AC5108696
Record Dates: First submitted 2007-11-06; First posted 2007-11-07 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Anticholinergic,; FTIH,; Muscarinic Receptor Antagonist,; Plethysmography; COPD,
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All subjects (Experimental): Eligible subjects will receive one of the following treatment in cohort I and cohort II in five different treatment periods; Placebo, GSK1160724 (10 micrograms, 50 micrograms or 125 micrograms) and tiotropium bromide
  Interventions: Drug: GSK1160724; Drug: Tiotropium bromide; Drug: Placebo

INTERVENTIONS:
Drug: GSK1160724 — GSK1160724 will be available with dosing strengths of 10, 50 and 125 micrograms/blister for inhalation using the DISKUS inhaler.
Drug: Tiotropium bromide — Tiotropium bromide capsules will be supplied with a dose of 18 micrograms administered via a HandiHaler device.
Drug: Placebo — Subjects will receive placebo.

SUMMARY:
GSK1160724 is a potent mAChR antagonist, which is being developed for treatment of chronic obstructive pulmonary disease (COPD)

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects. Female subjects must be of non-child bearing potential.
* Aged between 18-55 years inclusive
* Non-smokers
* Normal spirometry
* A signed and dated written informed consent is obtained from the subject
* The subject is capable of giving informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* Available to complete the study
* The subject is greater than or equal to 50kg with a body mass index within the range 19.0 to 29.9 kg/m2 inclusive
* Response to ipratropium bromide

Exclusion Criteria:

* Any clinically relevant and important abnormality identified at the screening medical assessment (physical examination/medical history), clinical laboratory tests, or ECG (12-lead or Holter)
* A history of breathing problems
* A mean QTc(B) value > 450ms, the QTc(B) of the 3 screening ECGs are not within 10% of the mean, a PR interval outside the range 90-210ms or an ECG that is not suitable for QT measurements at screening
* A history of elevated resting blood pressure or a mean blood pressure higher than 140/90 mmHg at screening
* A mean heart rate outside the range 40-90 bpm inclusive at screening
* History of use of tobacco- or nicotine-containing products within 6 months of screening, and/or positive urine cotinine test results at screening
* Where participation in the study would result in donation of blood in excess of 500mL within a 56 day period at screening
* The subject is currently taking regular (or a course of) medication, whether prescribed or not, including herbal remedies such as St John's Wort etc.

The subject has taken:

* prescription medications for 14 days prior to first dose of study drug, or
* Over-the-counter (OTC) medications/preparations (including herbal remedies, etc.) excluding simple analgesics for 48 hours prior to first dose of study drug,unless it is judged by the Investigator not to compromise the subject's safety or influence the outcome of the study.
* The subject has participated in a study with a new molecular entity or any other trial within a period of 3 months prior first dose of study drug
* The subject has tested positive for hepatitis C antibody (third generation enzyme immunoassay), hepatitis B surface antigen or HIV antibodies (if tested according to site SOP's) at screening.
* The subject has tested positive for drugs-of-abuse at screening
* The subject has tested positive for urine alcohol (including ethanol) at screening The detection of alcohol would not be an exclusion at screening but would need to be negative pre-dose and during the study
* The subject is unable to use the DISKUS™ and/or HandiHaler inhaler devices correctly at screening
* The subject has a suspected history of alcohol abuse within the six months previous to the screening visit
* The subject has a known allergy or hypersensitivity to magnesium stearate, milk protein or the excipient lactose monohydrate, iodine, ipratropium bromide, tiotropium bromide, atropine and/or any of its derivatives
* The subject has a significant clinical history of prostatic hypertrophy or narrow angle glaucoma
* The subject has received an allogeneic bone marrow transplant
* The subject has claustrophobia that may be aggravated by entering the whole body plethysmography cabinet

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2007-12-12 (Actual); Primary Completion 2008-04-07 (Actual); Study Completion 2008-04-07 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events (AEs) | Up to Week 24
  An AE is any untoward medical occurrence in a clinical study subjects, temporally associated with the use of a study treatment, whether or not considered related to the study treatment.
Number of subjects with abnormal values for blood pressure | Up to Week 24
  Systolic and diastolic blood pressure will be measured in a semi-recumbent position after 5 minutes rest.
Number of subjects with abnormal values for heart rate | Up to Week 24
  Heart rate will be measured in a semi-recumbent position after 5 minutes rest.
Number of subjects with abnormal electrocardiogram (ECG) findings | Up to Week 24
  Triplicate 12-lead ECGs will be measured in a semi-recumbent position after 5 minutes rest at each time point using ECG machine.
Number of subjects with abnormal findings after holter monitoring | Up to 24 hour
  Holter monitoring will be conducted at 24 hour.
Forced expiratory volume in 1 second (FEV1) | Up to Week 24
  Lung function will be measured by FEV1, defined as the maximal amount of air that can be forcefully exhaled in one second.
Forced vital capacity (FVC) | Up to Week 24
  Lung function will be measured by FVC, defined as the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible.
Number of subjects having abnormal hematology laboratory parameters | Up to Week 24
  Hematology parameters will be assessed as a measure of safety.
Number of subjects with abnormal clinical chemistry parameters | Up to Week 24
  Clinical parameters will be assessed as a measure of safety.
Number of subjects with abnormal values for urinalysis | Up to Week 24
  Urinalysis will be performed as a measure of safety.
Maximum value for resting heart rate over 0-4 hour | Up to 4 hours
  Maximum value for heart rate over 0-4 hour will be determined.
Maximum value for resting blood pressure over 0-4 hour | Up to 4 hours
  Maximum value for resting systolic and diastolic blood pressure over 0-4 hour will be determined.
Maximum value for resting ECG over 0-4 hour | Up to 4 hours
  Maximum value for resting ECG over 0-4 hour will be determined.
Weighted mean of resting heart rate over 0-4 hour | Up to 4 hours
  Weighted mean for resting heart rate over 0-4 hour will be determined.
Weighted mean of resting blood pressure over 0-4 hour | Up to 4 hours
  Weighted mean for resting systolic and diastolic blood pressure over 0-4 hour will be determined.
Weighted mean of resting ECG over 0-4 hour | Up to 4 hours
  Weighted mean for resting resting ECG over 0-4 hour will be determined.

SECONDARY OUTCOMES:
Plasma concentrations of GSK1160724 | Pre-dose, 5 minutes, 15 minutes, 30 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6 hours, 8 hours.12 hours, 16 hours, 24 hours, 48 hours Post-dose
  Plasma samples will be collected at the indicated time points to measure the concentration of GSK1160724.
Plasma concentrations of GSK1762245 | Pre-dose, 5 minutes, 15 minutes, 30 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6 hours, 8 hours.12 hours, 16 hours, 24 hours, 48 hours Post-dose
  Plasma samples will be collected at the indicated time points to measure the concentration of the active metabolite GSK1762245.
Urine concentrations of GSK1160724 | 0-2 hours, 2-8 hours, 8-12 hours and 12-24 hours
  Urine samples will be collected at the indicated time points to measure the concentration of GSK1160724.
Urine concentrations of GSK1762245 | 0-2 hours, 2-8 hours, 8-12 hours and 12-24 hours
  Urine samples will be collected at the indicated time points to measure the concentration of the active metabolite GSK1762245.
Maximum observed concentration (Cmax) of GSK1160724 | Pre-dose, 5 minutes, 15 minutes, 30 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6 hours, 8 hours.12 hours, 16 hours, 24 hours, 48 hours Post-dose
  Blood samples will be collected at the indicated time points for pharmacokinetic analysis.
Cmax of GSK1762245 | Pre-dose, 5 minutes, 15 minutes, 30 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6 hours, 8 hours.12 hours, 16 hours, 24 hours, 48 hours Post-dose
  Blood samples will be collected at the indicated time points for pharmacokinetic analysis.
Time to Cmax (Tmax) of GSK1160724 | Pre-dose, 5 minutes, 15 minutes, 30 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6 hours, 8 hours.12 hours, 16 hours, 24 hours, 48 hours Post-dose
  Blood samples will be collected at the indicated time points for pharmacokinetic analysis.
Tmax of GSK1762245 | Pre-dose, 5 minutes, 15 minutes, 30 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6 hours, 8 hours.12 hours, 16 hours, 24 hours, 48 hours Post-dose
  Blood samples will be collected at the indicated time points for pharmacokinetic analysis.
Time to last observed plasma concentration (Tlast) of GSK1160724 | Pre-dose, 5 minutes, 15 minutes, 30 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6 hours, 8 hours.12 hours, 16 hours, 24 hours, 48 hours Post-dose
  Blood samples will be collected at the indicated time points for pharmacokinetic analysis.
Tlast of GSK1762245 | Pre-dose, 5 minutes, 15 minutes, 30 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6 hours, 8 hours.12 hours, 16 hours, 24 hours, 48 hours Post-dose
  Blood samples will be collected at the indicated time points for pharmacokinetic analysis.
Area under the plasma concentration time curve from time 0 to last time of quantifiable concentration (AUC [0-T]) of GSK1160724 | Pre-dose, 5 minutes, 15 minutes, 30 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6 hours, 8 hours.12 hours, 16 hours, 24 hours, 48 hours Post-dose
  Blood samples will be collected at the indicated time points for pharmacokinetic analysis.
AUC (0-T) of GSK1762245 | Pre-dose, 5 minutes, 15 minutes, 30 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6 hours, 8 hours.12 hours, 16 hours, 24 hours, 48 hours Post-dose
  Blood samples will be collected at the indicated time points for pharmacokinetic analysis.
Area under the plasma concentration time curve from time 0 to infinity (AUC [0-infinity]) of GSK1160724 | Pre-dose, 5 minutes, 15 minutes, 30 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6 hours, 8 hours.12 hours, 16 hours, 24 hours, 48 hours Post-dose
  Blood samples will be collected at the indicated time points for pharmacokinetic analysis.
AUC (0-infinity) of GSK1762245 | Pre-dose, 5 minutes, 15 minutes, 30 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6 hours, 8 hours.12 hours, 16 hours, 24 hours, 48 hours Post-dose
  Blood samples will be collected at the indicated time points for pharmacokinetic analysis.
The terminal phase elimination rate constant (Lambda z) of GSK1160724 | Pre-dose, 5 minutes, 15 minutes, 30 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6 hours, 8 hours.12 hours, 16 hours, 24 hours, 48 hours Post-dose
  Blood samples will be collected at the indicated time points for pharmacokinetic analysis.
Lambda z of GSK1762245 | Pre-dose, 5 minutes, 15 minutes, 30 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6 hours, 8 hours.12 hours, 16 hours, 24 hours, 48 hours Post-dose
  Blood samples will be collected at the indicated time points for pharmacokinetic analysis.
The Terminal phase half life (T1/2) of GSK1160724 | Pre-dose, 5 minutes, 15 minutes, 30 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6 hours, 8 hours.12 hours, 16 hours, 24 hours, 48 hours Post-dose
  Blood samples will be collected at the indicated time points for pharmacokinetic analysis.
T1/2 of GSK1762245 | Pre-dose, 5 minutes, 15 minutes, 30 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6 hours, 8 hours.12 hours, 16 hours, 24 hours, 48 hours Post-dose
  Blood samples will be collected at the indicated time points for pharmacokinetic analysis.
Serial specific airway conductance (sGaw) response over 24 hours post-dose of GSK1160724 and tiotropium bromide | Up to 24 hours
  The sGaw response will be assessed by whole body plethysmograph at the indicated timepoints.
FEV1 over 24 hours post-dose of GSK1160724 and tiotropium bromide | Up to 24 hours
  The sGaw response will be assessed by whole body plethysmograph at the indicated timepoints.
FVC over 24 hours post-dose of GSK1160724 and tiotropium bromide | Up to 24 hours
  The sGaw response will be assessed by whole body plethysmograph at the indicated timepoints.
Serial sGaw measurements over 48 hours of GSK1160724 and tiotropium bromide | Up to 48 hours
  The sGaw is a measure of the change in specific airway conductance. It will be assessed by whole body plethysmograph at the indicated timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Harrow, Middlesex, United Kingdom

REFERENCES:
- See also: Results for study AC5108696 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/AC5108696?search=study&study_ids=AC5108696#rs